CLINICAL TRIAL: NCT05899855
Title: Foot Positions Affect Knee and Ankle Proprioception, Balance, Vertical Jump, and Muscle Activity in Individuals With Flexible and Rigid Flatfoot and Chronic Ankle Instability
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Ayman Mohamed, Beni-Suef University, Beni-Suef University
Other Study IDs: Cairo university
Record Dates: First submitted 2023-06-02; First posted 2023-06-12 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Flatfoot
MeSH Terms: conditions — Flatfoot

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: 30 subjects with rigid flatfoot and chronic ankle instability
  Interventions: Other: No intervention
- Group II: 30 subjects with flexible flatfoot and chronic ankle instability
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
To investigate the effect of various foot positions affect knee and ankle proprioception, balance, vertical jump, and muscle activity in individuals with flexible and rigid flatfoot and chronic ankle instability

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria were the presence of FF and chronic ankle instability in the dominant foot. Flexible and rigid flat feet were initially diagnosed by an orthopedist using a weight-bearing position with a standardized radiograph technique. The digital X-ray detector (film) and the X-ray tube (source) are 35-40 inches apart in lateral views of the foot. Then, Jack's test was performed to differentiate between the flexible and rigid FF. Jack's test is a valid test in assessing FF 10. Finally, people with flexible a second degree FF (Meary's angle between 15° to 30°) 3 were included in this study. The degree of flatfoot was determined by measuring the talus-first metatarsal angle on a lateral weight-bearing radiograph. This angle lies between a line drawn from the centers of the longitudinal axes of the talus and the first metatarsal. An angle that is greater than 4° convex downward is considered pes planus with an angle of 15° - 30° considered moderate, and greater than 30° severe 8. Chronic ankle instability was defined as the subject had a minimum of 2 acute ankle sprains, in the last 6 months, associated with pain, swelling, and a record of various ankle giving way. The determination of the dominant foot followed Vauhnik. & ark, modified version which stated that the dominant foot should be used minimally in 2 of the 3 subsequent activities: (1) Using the leg to step over a spider toy, (2) Drawing a diamond figure on the ground and (3) Kicking a ball.

Exclusion Criteria:

* The exclusion criteria were the existence of limited hallux dorsiflexion because Jack's test is valid only if hallux dorsiflexion is available during relaxed standing. Also, the participants were excluded if they had previous hip, pelvis, knee, or foot surgeries within the last year; obesity or pregnancy; leg-length discrepancies; has any vestibular disorder neurological disorder, brain concussion within the last 3 months that may cause balance impairment; or administering any drugs that could disturb alertness or balance.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Seventy-six participants met the inclusion and exclusion of this study. These participants were screened for the type of FF. We chose 30 for each group (60 total) to accomplish the balance between groups. Group 1: 30 subjects with rigid FF and chronic ankle instability, and Group 2: 30 subjects with flexible FF and chronic ankle instability. All participants were blinded to study procedures.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
knee proprioception | 2-3 months
  knee proprioception
ankle proprioception | 2-3 months
  ankle proprioception
Vertical jump measurements | 2-3 months
  Vertical jump measurements
Electromyographical activity (EMG) | 2-3 months
  Electromyographical activity (EMG)